CLINICAL TRIAL: NCT04290780
Title: Multicenter Study on Nosocomial Transmission of SARS-CoV-2 Virus
Brief Title: COVID-19 - Multicenter Study on Nosocomial Transmission of SARS-CoV-2 Virus
Acronym: NOSO-COR
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0214
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2022-01

CONDITIONS: Infection Viral
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — nasopharyngeal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: nosocomial infection/hospital acquired infection — When there is suspicion of a community-acquired case (admission of an infected patient) or nosocomial case (infection of a patient already hospitalized), a case report form including demographic data, medical history, and clinical and biological data on the infectious episode will be completed for each case, either patient, caregivers or health care professionals, presenting clinical signs or symptoms compatible with SARS-CoV-2 infection. The suspected cases will undergo nasopharyngeal swab collection and detection of SARS-CoV-2 in nasopharyngeal swabs will be done by real-time RT-PCR assay.
  Hygiene measures applied by the service will be collected using a questionnaire as well as recommendations of the learned societies within the country regarding the risk of infection by coronavirus. In addition, data characterizing the service and hospital will also be collected (specialty, number of beds, number of nurses, doctors, etc.).

SUMMARY:
Infection with the SARS-CoV-2 coronavirus strain is associated with severe morbidity and mortality estimated today from 2% to 4%. Elderly patients or patients with serious chronic conditions justifying hospitalization are particularly at risk. The risk of infection with SARS-CoV-2 during hospitalization is also substantial and increased in fragile patients. Several cases of infection among Healthcare Professionals had been reported.

The hypothesis is that similar to the corona virus agent responsible for SRAS and the influenza virus, nosocomial outbreaks of SARS-CoV-2 to be feared. Health care professionals and caregivers are populations-at-risk as they are exposed in the community and can transmit SARS-CoV-2 to hospitalized patients, and are also exposed to hospitalized patients infected with SARS-CoV-2.

Describing hospital-acquired cases and SARS-CoV-2 infection transmission chains in healthcare settings is vitally essential to achieve control of this epidemic. To improve the quality of care and patient safety, this data must be accompanied by an analysis of the impact of infection control measures. In addition, an effective infection control program is urgently required to control the spread of the virus and protect both uninfected patients who require care for other medical or surgical conditions as well as health care professionals.

The main objective of this prospective, non-interventional - observational, hospital based study in adults and children is to describe and document suspected or confirmed cases of nosocomial SARS-CoV-2 infection, the clinical spectrum and the determinants (risk factors/protective factors) at participating hospitals.

Characterization of the clinical features of the SARS-CoV-2 infection will help to identify potential sources of virus transmission as rapidly as possible and enable implementation of appropriate hygiene practices in hospitals.

ELIGIBILITY:
Inclusion Criteria:

1 ) Any adult or child or member of the nursing staff from the study participant hospital who presents an infectious syndrome including the following definition :

2) Suspect Case:

Fever above 37.8 ° C if no antipyretics are taken; And or Cough or pharyngeal pain or other symptom suggestive of respiratory infection. AND at least 1 of the following characteristics:

* return from a trip to China, or to a country in which the increase in the incidence of infections in SARS-CoV-2 has been proven;
* close contact (sharing the same place of family, professional life, same plane, etc.) with a person defined as a suspected or confirmed case;
* Occurring in an establishment having received at least one case of suspected or confirmed infection at SARS-CoV-2.

Or 3) Confirmed Case: The same clinical definitions, in addition to a positive RT-PCR-type virological diagnostic result specific to SARS-CoV-2

Exclusion Criteria:

* Anyone who does not meet the above definition.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will focus on volunteers, patients, caregivers and health care professionals within the participating hospitals associated with the GABRIEL network. Other hospitals, including french, will be able to integrate with this project on a voluntary basis.
Sampling Method: Non-Probability Sample
Enrollment: 2162 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
nosocomial infection | At inclusion
  The primary outcome criteria will be the proportion of patients, caregivers and health care professionals with confirmed or suspected SARS-CoV-2 nosocomial infection relative to all patients, caregivers and health care professionals with syndromes suggestive of SARS-CoV-2 infection during the study period. The infection control measures will be reported and describe according the nosocomial cases.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe VANHEMS, MD, PhD, Principal Investigator — Service Hygiène, Epidémiologie et Prévention
Locations (1):
- Service Hygiène, Epidémiologie et Prévention, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saadatian-Elahi M, Picot V, Henaff L, Pradel FK, Escuret V, Dananche C, Elias C, Endtz HP, Vanhems P. Protocol for a prospective, observational, hospital-based multicentre study of nosocomial SARS-CoV-2 transmission: NOSO-COR Project. BMJ Open. 2020 Oct 22;10(10):e039088. doi: 10.1136/bmjopen-2020-039088. PMID 33093033
- [Derived] Vanhems P. A breath of humanity in the era of Covid-19 vaccine. Vaccine. 2021 Jun 23;39(28):3649. doi: 10.1016/j.vaccine.2021.05.052. Epub 2021 May 24. No abstract available. PMID 34053788